CLINICAL TRIAL: NCT01980069
Title: A Double-blind, Randomized, Parallel Design Study to Compare the Effectiveness of Sugammadex Versus Neostigmine in Improving Surgical Condition in Subjects Undergoing Laryngeal Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0451
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: General Anesthesia
Keywords: Sugammadex; Neostigmine; Surgery
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neostigmine arm (Experimental): Neostigmine arm
  Interventions: Drug: Neostigmine
- Sugammadex arm (Active Comparator): Sugammadex arm
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — In sugammadex group, sugammadex (Bridion, Merck Shart and Dohme (MSD), Oss, the Netherlands) will be administered intravenously in different doses according to the degree of muscle relaxation. Sugammadex 8 mg/kg will be administered if there is no response on post-tetanic count (PTC) stimulus. Sugammadex 4 mg/kg will be administered if PTC is more than 1 or 2. Sugammadex 2 mg/kg will be administered if T2 response appears on train-of-four (TOF) stimulus.
  Arms: Sugammadex arm
Drug: Neostigmine — In neostigmine group, neostigmine 50 ㎍/kg will be administered intravenously with glycopyrrolate 10 ㎍/kg when the T2 response appears on TOF stimuli.
  Arms: Neostigmine arm

SUMMARY:
Investigators hypothesized that the surgical condition will be improved with the use of sugammadex in patients undergoing laryngeal microsurgery. Investigators will compare the effect of sugammadex and neostigmine on the surgical condition during laryngeal microsurgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of age over 20 years
* scheduled for laryngeal microsurgery under general anesthesia

Exclusion Criteria:

* anticipated difficult intubation, cervical spine disease, neuromuscular disease, acute or chronic renal failure, liver cirrhosis or liver failure
* history of allergy to nondepolarizing muscle relaxant
* history of malignant hyperthermia
* pregnant woman
* body mass index over 35 kg/m2

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
surgical condition | up to 1 hour after the end of surgery
  Primary outcome is the proportion of patients who have clinically acceptable surgical condition. The surgeon will evaluate the surgical condition as a surgical rating scale during surgery (extremely poor condition, poor condition, acceptable condition, good condition, optimal condition).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

REFERENCES:
- [Derived] Kim HJ, Lee K, Park WK, Lee BR, Joo HM, Koh YW, Seo YW, Kim WS, Yoo YC. Deep neuromuscular block improves the surgical conditions for laryngeal microsurgery. Br J Anaesth. 2015 Dec;115(6):867-72. doi: 10.1093/bja/aev368. PMID 26582847